CLINICAL TRIAL: NCT00497913
Title: Dysport® Injection in the Treatment of Chronic Lateral Epicondylitis
Acronym: DCLE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 85-02-53-4207
Record Dates: First submitted 2007-07-06; First posted 2007-07-09 (Estimated); Last update posted 2008-04-23 (Estimated); Status verified 2008-04

CONDITIONS: Tennis Elbow
Keywords: Tennis Elbow; Botulinum Toxin
MeSH Terms: conditions — Tennis Elbow | interventions — Sodium Chloride; Botulinum Toxins, Type A; abobotulinumtoxinA

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: Botulinum Toxin A
- B (Placebo Comparator)
  Interventions: Drug: NaCl 0.9%

INTERVENTIONS:
Drug: NaCl 0.9%
  Arms: B
Drug: Botulinum Toxin A
  Other Names: Dysport
  Arms: A

SUMMARY:
The purpose of this study is to determine whether a single injection of Dysport with a new protocol at forearm is effective in the management of chronic lateral epicondylitis.

DETAILED DESCRIPTION:
Some studies valued the effectiveness of botulinum toxin. There is a great amount of controversy on the amount of botulinum toxin injected and the location of the injection. The purpose of the study is to compare the effectiveness of botulinum toxin injection with placebo at a new injection site at the forearm in the treatment of chronic tennis elbow unrelieved by corticosteroid injection and physiotherapy. It is a double blind randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Pain: pain will be assessed as the physician touches lateral epicondyle or passively flexing the patient's wrist and while the patient extends his/her wrist or 3rd finger against resistance. Individuals who fulfill two or more of above will be considered to have lateral epicondylitis.
* Symptom duration: should be at least 6 months.
* Previous trial of complete course of physiotherapy and corticosteroid injection.

Exclusion Criteria:

* Rheumatoid arthritis
* Generalized polyarthritis
* Local elbow arthritis
* Simultaneous medial epicondylalgia
* Bilateral lateral epicondylitis
* Neurologic deficits (abnormal light touch sensation, deep tendon reflexes abnormality, radicular pain, radial nerve entrapment, signs of nerve root compression, decreased muscle force, multiple sclerosis, seizures)
* The use of corticosteroid in last 30 days
* Simultaneous use of drugs other than acetaminophen or physical therapy in the course of study
* Pregnancy
* Breast-feeding
* Previous hand surgery
* Having a hobby or job that needs finger extension

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2007-08; Primary Completion 2008-03 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Pain score on VAS at maximal grip, at maximal pinch, and during previous month at rest | 4 months

SECONDARY OUTCOMES:
Patients subjective feeling of improvement. | 4 months
Tenderness on lateral epicondyle | 4 months
Pain sensation on resisted wrist extension, and passive wrist flexion | 4 months
Pain-free grip strength, and pinch strength | 4 months
Maximal grip strength, and pinch strength | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Seyed Mohammad J Mortazavi, M.D., Study Director — Tehran University of Medical Sciences
Locations (1):
- Imam Khomeini Hospital, Tehran, Tehran Province, Iran

REFERENCES:
- [Derived] Espandar R, Heidari P, Rasouli MR, Saadat S, Farzan M, Rostami M, Yazdanian S, Mortazavi SM. Use of anatomic measurement to guide injection of botulinum toxin for the management of chronic lateral epicondylitis: a randomized controlled trial. CMAJ. 2010 May 18;182(8):768-73. doi: 10.1503/cmaj.090906. Epub 2010 Apr 26. PMID 20421357